CLINICAL TRIAL: NCT01841957
Title: Immediate Simultaneous Bilateral Cataract Surgery: A Prospective, Case-controlled Clinical Trial in the United States
Brief Title: Immediate Simultaneous Bilateral Cataract Surgery
Acronym: ISBCS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sloan W. Rush, MD (Other)
Responsible Party: Sponsor-Investigator, Sloan W. Rush, MD, MD, Panhandle Eye Group, LLP
Organization: Panhandle Eye Group, LLP (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2
Record Dates: First submitted 2013-04-18; First posted 2013-04-29 (Estimated); Last update posted 2022-04-28 (Actual); Status verified 2022-04

CONDITIONS: Bilateral Cataract
Keywords: Bilateral Cataract; Simultaneous Cataract Surgery; ISBCS
MeSH Terms: conditions — Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- ISBCS (Experimental): Immediate Simultaneous Bilateral Cataract Surgery
  Interventions: Procedure: ISBCS
- DSBCS (Active Comparator): Delayed Sequential Bilateral Cataract Surgery
  Interventions: Procedure: DSBCS

INTERVENTIONS:
Procedure: ISBCS — same-day cataract surgery
  Arms: ISBCS
Procedure: DSBCS — bilateral surgery delayed by 1-3 weeks amongst eyes
  Arms: DSBCS

SUMMARY:
To evaluate the safety and efficacy of treating visually significant bilateral cataract with the newer technique of Immediate Simultaneous Bilateral Cataract Surgery (ISBCS) versus the conventional technique of Delayed Sequential Bilateral Cataract Surgery (DSBCS) in a select patient population.

ELIGIBILITY:
Inclusion Criteria:

* Age 30-100
* Candidate for topical anesthesia
* Signed the informed consents

Exclusion Criteria:

* Allergies to medications used in study
* Cannot have topical anesthesia
* Unwilling to participate in research trial
* Have any other significant ocular comorbidities
* Have known systemic immuno-compromised state

Ages: 30 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-04 (Actual); Primary Completion 2022-04-01 (Actual); Study Completion 2022-04-01 (Actual)

PRIMARY OUTCOMES:
Visual acuity | 3 weeks
  Best uncorrected and best spectacle corrected post-operative visual acuity

SECONDARY OUTCOMES:
Recovery time and number of post-operative visits | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Panhandle Eye Group, Amarillo, Texas, United States